CLINICAL TRIAL: NCT04619563
Title: A Single-arm Exploratory Clinical Study of Anlotinib Hydrochloride Combined With Docetaxel in EGFR Mutations Advanced Non Small Cell Lung Cancer Patients Who Have Progressed After Targeted Therapy and Chemotherapy
Brief Title: A Trial of Anlotinib Combined With Docetaxel in EGFR Mutations Advanced Non Small Cell Lung Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jinming Yu, President of Shandong Cancer Hospital and Institute, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2020-052-02
Record Dates: First submitted 2020-11-03; First posted 2020-11-06 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Anlotinib Hydrochloride; Docetaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib hydrochloride plus Docetaxel (Experimental): Paticipants receive 4 to 6 cycles (21 days per cycle) combined administration period of Anlotinib Hydrochloride and Docetaxel, and then Anlotinib Hydrochloride maintenance treatment.
  Interventions: Drug: Anlotinib Hydrochloride plus Docetaxel

INTERVENTIONS:
Drug: Anlotinib Hydrochloride plus Docetaxel — Anlotinib Hydrochloride (12mg, QD PO d1-14, 21days per cycle) and Docetaxel (75mg/m2 IV d1)
  Other Names: Fu Ke Wei

SUMMARY:
Anlotinib is a multi-target receptor tyrosine kinase inhibitor in domestic research and development. It can inhibit angiogenesis-related kinases, such as VEGFR, FGFR, PDGFR and tumor cell proliferation related kinase c-Kit kinase. In the Phase III study, patients who failed at least two systemic chemotherapy (third-line or above) or were intolerant of the drugs were treated with anlotinib or placebo. The PFS and OS in the anlotinib group were 5.37 months and 9.63 months, respectively. The placebo group PFS and OS were 1.4 months and 6.3 months. Therefore, it is envisaged to use anlotinib combined with docetaxel to treat EGFR mutations advanced non small cell lung cancer to further improve the patient's PFS or OS.

DETAILED DESCRIPTION:
This is a single arm clinical trial conducted in China. The purpose of this study is to evaluate and observe the efficacy and safety of Anlotinib Hydrochloride (12mg, QD PO d1-14, 21days per cycle) combined with Docetaxel (75mg/m2 IV d1) in EGFR mutations advanced non small cell lung cancer patients who have progressed after targeted therapy and chemotherapy. After being informed about the study and potential risks, all patients giving written informed consent will undergo a 4-week screening period to determine eligibility for study entry. The expected sample size is 42.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily join the study and sign an informed consent form, with good compliance and cooperation with follow-up.
* EGFR mutation-positive、ALK mutation-negative；Patients have progressed after receiving EGFR targeted and chemotherapy as first-line treatment.
* Patients who were resistant to EGFR targeted treatment need to receive T790M mutation test. If the test is positive and Patients have not orally taken osimertinib or almonertinib, patients need to orally taken osimertinib or almonertinib and be progressed prior to enrollment.
* ≥ 18 and ≤ 75 years of age; female or male.
* Diagnosed with local advanced and/or metastatic NSCLC (phase IIIB、IIIC or IV) through Histology or cytology (using the new version of staging announced by the American Joint Committee on Cancer on January 1, 2018), or recurrent non- squamous non-small cell lung cancer. Noted: failed from prior treatment means(1) progress disease confirmed by definite imageology and clinical evidence during treatment or after the last treatment; (2) Patients withdrew from treatment because of intolerant adverse events, the intolerant adverse events refer to≥ level IV hematologic toxicities or ≥ level III non-hematologic toxicities or ≥ level 2 damages of major organs such as heart/liver/kidney in CTC AE 4.0.
* There is at least one target lesion that has not received radiotherapy, and it can be accurately measured by magnetic resonance imaging (MRI) or computed tomography (CT) in at least one direction (the maximum diameter needs to be recorded), where the maximum tumor diameter is >10 mm; the shortest diameter of the lymph node is >15mm.
* Expected survival time: at least 3 months
* ECOG PS：0-1
* The damage caused by other treatments has been recovered (NCI-CTCAE 4.0 version classification≤level 1); Radiotherapy (except local palliative radiotherapy)≥ 2 weeks.
* The main organs function are normally, the following criteria are met

  1. Blood routine examination criteria should be met (no blood transfusion and blood products within 14 days): HB≥90 g/L; ANC ≥ 1.5×10^9/L; PLT ≥80×10^9/L;
  2. Biochemical examinations must meet the following criteria: TBIL<1.5ULN; ALT and AST < 2.5ULN, and for patients with liver metastases < 5ULN; Serum Cr ≤ 1.25ULN or endogenous creatinine clearance > 45ml/min (Cockcroft-Gault formula);
* Women of childbearing potential must have taken reliable contraceptive measures or the result of serum or urine pregnancy test should be negative within 7 days prior to study enrollment, and willing to use and utilize an adequate method of contraception throughout treatment and for at least 8 weeks after the last test drug administration. Man participants should agree to use and utilize an adequate method of contraception throughout treatment and for at least 8 weeks after the last test drug administration or surgical sterilization.

Exclusion Criteria:

* Squamous carcinoma of lung (including Adenosquamous carcinoma); Small cell lung cancer (including lung cancer mixed with small cell lung cancer and non- small cell lung cancer);
* Have used Anlotinib Hydrochloride、docetaxel before; Postoperative adjuvant therapy with docetaxel is acceptable.
* Imaging (CT or MRI) shows that the distance between tumor lesion and the large blood vessel is ≤ 5 mm, or there is a central tumor that invades the local large blood vessel; or there is a significant pulmonary cavity or necrotizing tumor;
* Medical history and combined history：

  1. Significant brain metastases, cancerous meningitis, spinal cord compression, or imaging CT or MRI screening for brain or pia mater disease (a patient with brain metastases who have completed treatment and stable symptoms in 28 days before enrollment may be enrolled, but should be confirmed by brain MRI, CT or venography evaluation as no cerebral hemorrhage symptoms);
  2. The patient is participating in other clinical studies.
  3. Other active malignancies that require simultaneous treatment;
  4. Patients with a history of malignant tumors except for patients with cutaneous basal cell carcinoma, superficial bladder cancer, cutaneous squamous cell carcinoma or orthotopic cervical cancer who have undergone a possible curative treatment and have no disease recurrence within 5 years from the start of treatment;
  5. Patients with previously systemic anti-tumor treatment-related adverse reactions (excluding hair loss) who have not recovered to NCI-CTCAE ≤level 1;
  6. Abnormal blood coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT > 1.5 ULN), with bleeding tendency or undergoing thrombolytic or anticoagulant therapy; Note: Under the premise of prothrombin time international normalized ratio (INR) ≤ 1.5, low-dose heparin (adult daily dose of 0.6 million to 12,000 U) or low-dose aspirin (daily dosage ≤ 100 mg) is allowed for preventive purposes;
  7. Renal insufficiency: urine routine indicates urinary protein ≥ ++, or confirmed 24-hour urine protein ≥ 1.0g;
  8. The effects of surgery or trauma have been eliminated for less than 14 days before enrollment in subjects who have undergone major surgery or have severe trauma;
  9. Severe acute or chronic infections requiring systemic treatment;
  10. Suffering from severe cardiovascular disease: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmias (including men with QTc interval ≥ 450 ms, women ≥ 470 ms); according to NYHA criteria, grades III to IV Insufficient function, or cardiac color Doppler ultrasound examination indicates left ventricular ejection fraction (LVEF) <50%;
  11. Peripheral neuropathy with ≥CTCAE degree 2 currently exists, except for trauma caused;
  12. Respiratory syndrome (≥CTC AE grade 2 dyspnea), serous effusion (including pleural effusion, ascites, pericardial effusion) requiring treatment;
  13. Long-term unhealed wounds or fractures;
  14. Decompensated diabetes or other ailments treated with high doses of glucocorticoids;
  15. Factors that have a significant impact on oral drug absorption, such as inability to swallow, chronic diarrhea, and intestinal obstruction;
  16. Clinically significant hemoptysis (daily hemoptysis greater than 50ml) within 3 months before enrollment; or significant clinically bleeding symptoms or defined bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood ++ and above, or suffering from vasculitis;
  17. Events of arterious/venous thrombosis occurring within 12 months prior to enrollment, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
  18. Planned for systemic anti-tumor therapy, including cytotoxic therapy, signal transduction inhibitors, immunotherapy. Extended-field radiotherapy (EF-RT) was performed within 3 weeks before grouping or limited-field radiotherapy to be evaluated for tumor lesions within 2 weeks before grouping;
  19. Uncontrollable hypertension with two or more combined treatments (systolic blood pressure ≥145 mmHg or diastolic blood pressure ≥90 mmHg);
  20. Have a history of psychotropic substance abuse and are unable to quit or have a mental disorder;
* Physical examination and laboratory examination findings

  1. A known history of HIV testing positive or acquired immunodeficiency syndrome (AIDS);
  2. untreated active hepatitis (hepatitis b: HBsAg positive and HBV DNA ≥500 IU/ml; Hepatitis c: HCV RNA is positive and liver function is abnormal); Combined with hepatitis b and hepatitis c infection;
* Other factors that may cause the study to be terminated midway according to the researchers' judgment, such as other serious diseases or severe laboratory test abnormalities or factors that will endanger patients' safety, or family or society factors of test data and sample collection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Progress free survival (PFS) | each 42 days up to PD or death (up to 24 months)
  PFS is defined as the time from the date of enrollment to the first occurrence of disease progression or death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.prior to progression or any further therapy.
Disease Control Rate (DCR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  DCR is defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1.
Overall Survival (OS) | From randomization until death (up to 24 months)
  OS is defined as the time from the date of enrollment to the date of death due to any cause.
Quality of Life score (QoL) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  use EORTC QLQ-C30(version 3) questionnaire to evaluate the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Cancer Hospital, Jinan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Background] Park K, Tan EH, O'Byrne K, Zhang L, Boyer M, Mok T, Hirsh V, Yang JC, Lee KH, Lu S, Shi Y, Kim SW, Laskin J, Kim DW, Arvis CD, Kolbeck K, Laurie SA, Tsai CM, Shahidi M, Kim M, Massey D, Zazulina V, Paz-Ares L. Afatinib versus gefitinib as first-line treatment of patients with EGFR mutation-positive non-small-cell lung cancer (LUX-Lung 7): a phase 2B, open-label, randomised controlled trial. Lancet Oncol. 2016 May;17(5):577-89. doi: 10.1016/S1470-2045(16)30033-X. Epub 2016 Apr 12. PMID 27083334
- [Background] Wu YL, Cheng Y, Zhou X, Lee KH, Nakagawa K, Niho S, Tsuji F, Linke R, Rosell R, Corral J, Migliorino MR, Pluzanski A, Sbar EI, Wang T, White JL, Nadanaciva S, Sandin R, Mok TS. Dacomitinib versus gefitinib as first-line treatment for patients with EGFR-mutation-positive non-small-cell lung cancer (ARCHER 1050): a randomised, open-label, phase 3 trial. Lancet Oncol. 2017 Nov;18(11):1454-1466. doi: 10.1016/S1470-2045(17)30608-3. Epub 2017 Sep 25. PMID 28958502
- [Background] Mok TS, Wu Y-L, Ahn M-J, Garassino MC, Kim HR, Ramalingam SS, Shepherd FA, He Y, Akamatsu H, Theelen WS, Lee CK, Sebastian M, Templeton A, Mann H, Marotti M, Ghiorghiu S, Papadimitrakopoulou VA; AURA3 Investigators. Osimertinib or Platinum-Pemetrexed in EGFR T790M-Positive Lung Cancer. N Engl J Med. 2017 Feb 16;376(7):629-640. doi: 10.1056/NEJMoa1612674. Epub 2016 Dec 6. PMID 27959700
- [Background] Soria JC, Ohe Y, Vansteenkiste J, Reungwetwattana T, Chewaskulyong B, Lee KH, Dechaphunkul A, Imamura F, Nogami N, Kurata T, Okamoto I, Zhou C, Cho BC, Cheng Y, Cho EK, Voon PJ, Planchard D, Su WC, Gray JE, Lee SM, Hodge R, Marotti M, Rukazenkov Y, Ramalingam SS; FLAURA Investigators. Osimertinib in Untreated EGFR-Mutated Advanced Non-Small-Cell Lung Cancer. N Engl J Med. 2018 Jan 11;378(2):113-125. doi: 10.1056/NEJMoa1713137. Epub 2017 Nov 18. PMID 29151359
- [Background] Han B, Li K, Wang Q, Zhang L, Shi J, Wang Z, Cheng Y, He J, Shi Y, Zhao Y, Yu H, Zhao Y, Chen W, Luo Y, Wu L, Wang X, Pirker R, Nan K, Jin F, Dong J, Li B, Sun Y. Effect of Anlotinib as a Third-Line or Further Treatment on Overall Survival of Patients With Advanced Non-Small Cell Lung Cancer: The ALTER 0303 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2018 Nov 1;4(11):1569-1575. doi: 10.1001/jamaoncol.2018.3039. PMID 30098152